CLINICAL TRIAL: NCT01212666
Title: The Effect of Adductor-Canal-Block (ACB) in Patients After Anterior Cruciate Ligament (ACL) Reconstruction in Day Case Surgery
Brief Title: The Efficacy of Adductor-Canal-Block (ACB) in Patients After Anterior Cruciate Ligament (ACL) Reconstruction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, Malene Espelund, MD, Glostrup University Hospital, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SM1-ME-10
Record Dates: First submitted 2010-05-26; First posted 2010-10-01 (Estimated); Last update posted 2012-09-11 (Estimated); Status verified 2012-09

CONDITIONS: Anterior Cruciate Ligament Reconstruction
Keywords: Adductor Canal Block (ACB); Anterior Cruciate Ligament (ACL) Reconstruction; Saphenous nerve; Pain; Ultrasound block
MeSH Terms: conditions — Pain | interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adductor-Canal-Block, Ropivacain (Experimental): 25 patients. ACB. 30 mL Ropivacain 7,5 mg/mL. Ultrasound-guided application.
  Interventions: Procedure: Ropivacain
- Adductor Canal Block, Placebo (saline) (Placebo Comparator): 25 patients. ACB. 30 mL Saline. Ultrasound-guided application.
  Interventions: Procedure: Saline

INTERVENTIONS:
Procedure: Ropivacain — Ultrasound-guided ACB; 30 mL Ropivacain 7,5 mg/mL. Single dose.
  Other Names: Naropin
  Arms: Adductor-Canal-Block, Ropivacain
Procedure: Saline — Ultrasound-guided Adductor Canal Block; 30 mL Saline. Single dose.
  Arms: Adductor Canal Block, Placebo (saline)

SUMMARY:
The Purpose of this study is to determine whether Adductor-Canal-Block is superior to placebo when it comes to analgetic efficacy after reconstruction of the anterior cruciate ligament.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years
* Reconstruction of Anterior Cruciate Ligament
* Written consent
* ASA I-II
* BMI 19-35

Exclusion Criteria:

* Unable to communicate in Danish
* Allergic reactions toward drugs used in the trial
* Pregnancy
* Abuse of alcohol/drugs
* Daily opioid intake
* Infection at injection site
* Can not be mobilised to 5 meters of walk; pre-surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-05; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Pain-score (VAS), patient standing | 2 hours postoperative
  Pain-score messured on a Visual Analog Scale (VAS) 2 hours after adductor canal block. Patient standing. Intervention-group vs. placebo-group.

SECONDARY OUTCOMES:
Total Opioid-consumption | 0-24 hours postoperative
  ACB-group vs. placebo-group
Postoperative Nausea and Vomiting | 0 hour postoperative
  Levels of nausea (0-3). ACB-group vs. placebo-group
Postoperative ondansetron consumption | In hospital
Pain-score (VAS), patient at rest | 0 hours postoperative
  ACB-group vs. placebo
Pain-score (VAS), patient at rest | 1 hour postoperative
  ACB-group vs. placebo
Pain-score (VAS), patient at rest | 2 hours postoperative
  ACB-group vs. placebo
Pain-score (VAS), patient at rest | 4 hours postoperative
  ACB-group vs. placebo
Pain-score (VAS), patient at rest | 6 hours postoperative
  ACB-group vs. placebo
Pain-score (VAS), patient at rest | 8 hours postoperative
  ACB-group vs. placebo
Pain-score (VAS), patient at rest | 24 hours postoperative
  ACB-group vs. placebo
Pain-score (VAS), patient standing | 1 hour postoperative
  ACB-group vs. placebo
Pain-score (VAS), patient standing | 2 hours postoperative
  ACB-group vs. placebo
Pain-score (VAS), patient standing | 4 hours postoperative
  ACB-group vs. placebo
Pain-score (VAS), patient standing | 6 hours postoperative
  ACB-group vs. placebo
Pain-score (VAS), patient standing | 8 hours postoperative
  ACB-group vs. placebo
Pain-score (VAS), patient standing | 24 hours postoperative
  ACB-group vs. placebo
Pain-score (VAS), after 5 meters of walk | 2 hours postoperative
  ACB-group vs. placebo
Pain-score (VAS), after 5 meters of walk | 4 hours postoperative
  ACB-group vs. placebo
Pain-score (VAS), after 5 meters of walk | 6 hours postoperative
  ACB-group vs. placebo
Pain-score (VAS), after 5 meters of walk | 8 hours postoperative
  ACB-group vs. placebo
Pain-score (VAS), after 5 meters of walk | 24 hours postoperative
  ACB-group vs. placebo
Postoperative Nausea and Vomiting | 1 hours postoperative
  Levels of nausea (0-3). ACB-group vs. placebo-group
Postoperative Nausea and Vomiting | 2 hours postoperative
  Levels of nausea (0-3). ACB-group vs. placebo-group
Postoperative Nausea and Vomiting | 4 hours postoperative
  Levels of nausea (0-3). ACB-group vs. placebo-group
Postoperative Nausea and Vomiting | 6 hours postoperative
  Levels of nausea (0-3). ACB-group vs. placebo-group
Postoperative Nausea and Vomiting | 8 hours postoperative
  Levels of nausea (0-3). ACB-group vs. placebo-group
Postoperative Nausea and Vomiting | 24 hours postoperative
  Levels of nausea (0-3). ACB-group vs. placebo-group
Sedation | 0, hour postoperative
  Levels of sedation (0-3). ACB-group vs. placebo
Sedation | 1 hour postoperative
  Levels of sedation (0-3). ACB-group vs. placebo
Sedation | 2 hours postoperative
  Levels of sedation (0-3). ACB-group vs. placebo
Sedation | 4 hours postoperative
  Levels of sedation (0-3). ACB-group vs. placebo
Sedation | 6 hours postoperative
  Levels of sedation (0-3). ACB-group vs. placebo
Sedation | 8 hours postoperative
  Levels of sedation (0-3). ACB-group vs. placebo
Sedation | 24 hours postoperative
  Levels of sedation (0-3). ACB-group vs. placebo
Postoperative Nausea and Vomiting | 0 hours postoperative
  Levels of nausea (0-3). ACB-group vs. placebo-group
Pain (VAS) at rest, 0-24 hours postoperative (AUC) | 0-24 h postoperative
  Pain-score messured on a Visual Analog Scale (VAS) 0-24 hours after adductor canal block (AUC). Patient at rest. Intervention-group vs. placebo-group.
Pain (VAS), patient standing, 1-24 hours postoperative (AUC) | 1-24 hours postoperative
  Pain-score messured on a Visual Analog Scale (VAS) 1-24 hours after adductor canal block (AUC). Patient standing. Intervention-group vs. placebo-group.
Pain (VAS), pain after 5 meters of walk, 2-24 hours postoperative (AUC) | 2-24 hours postoperative
  Pain-score messured on a Visual Analog Scale (VAS) 2-24 hours after adductor canal block (AUC). Pain after 5 meters of walk. Intervention-group vs. placebo-group.

CONTACTS AND LOCATIONS:
Overall Officials: Malene Espelund, MD, Principal Investigator — Glostrup University Hospital, Copenhagen
Locations (1):
- Department of Anaesthesiology, Glostrup University Hospital, Copenhagen, Glostrup, Denmark

REFERENCES:
- [Derived] Espelund M, Fomsgaard JS, Haraszuk J, Mathiesen O, Dahl JB. Analgesic efficacy of ultrasound-guided adductor canal blockade after arthroscopic anterior cruciate ligament reconstruction: a randomised controlled trial. Eur J Anaesthesiol. 2013 Jul;30(7):422-8. doi: 10.1097/EJA.0b013e328360bdb9. PMID 23549123